CLINICAL TRIAL: NCT06268613
Title: A Phase I, Randomised, Double-blind, Three-arm, Parallel Group, Multicentre Study to Compare the Pharmacokinetics (PK), Efficacy, Safety, and Immunogenicity of Pembrolizumab (SB27, European Union [EU] Sourced Keytruda, and the United States of America [US] Sourced Keytruda) in Subjects With Stage II-IIIA Non-small Cell Lung Cancer Following Complete Resection and Adjuvant Platinum-based Chemotherapy
Brief Title: A Study to Compare the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of Pembrolizumab (SB27, EU Sourced Keytruda, and US Sourced Keytruda) in Subjects With Stage II-IIIA NSCLC Following Complete Resection and Adjuvant Platinum-based Chemotherapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB27-1005
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage IIIA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SB27 (Experimental): SB27 will be administered intravenously at a fixed dose of 200 mg every 3 weeks, maximum 18 cycles over about 51 weeks
  Interventions: Drug: SB27
- EU sourced Keytruda (Active Comparator): EU sourced Keytruda will be administered intravenously at a fixed dose of 200 mg every 3 weeks, maximum 18 cycles over about 51 weeks
  Interventions: Drug: EU sourced Keytruda
- US sourced Keytruda (Active Comparator): EU sourced Keytruda will be administered intravenously at a fixed dose of 200 mg every 3 weeks, maximum 18 cycles over about 51 weeks
  Interventions: Drug: US sourced Keytruda

INTERVENTIONS:
Drug: SB27 — Will be administered intravenously at a fixed dose of 200 mg every 3 weeks, maximum 18 cycles over about 51 weeks
  Arms: SB27
Drug: EU sourced Keytruda — Will be administered intravenously at a fixed dose of 200 mg every 3 weeks, maximum 18 cycles over about 51 weeks
  Arms: EU sourced Keytruda
Drug: US sourced Keytruda — Will be administered intravenously at a fixed dose of 200 mg every 3 weeks, maximum 18 cycles over about 51 weeks
  Arms: US sourced Keytruda

SUMMARY:
The goal of this clinical trial is to compare the amount of study drug in patients' blood to confirm that SB27 works in the same way as EU and US sourced Keytruda in early or locally advanced non-small cell lung cancer (NSCLC) patients who underwent surgery and adjuvant chemotherapy. The main question it aims to answer is:

• What the body does to the study drug, which is called "pharmacokinetic"

Participants will receive investigational product (IP) administration every 3 weeks, maximum 18 cycles over about 51 weeks and blood sample will be collected.

Researchers will compare 3 medicines (SB27, EU sourced Keytruda, and US sourced Keytruda) to see if SB27 works in the same way as EU and US sourced Keytruda.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Diagnosed as NSCLC stage II-IIIA (staging should be confirmed after surgery)
* Have completely removed all of the cancer from the body surgically
* Have been received 3 or 4 cycles of platinum-based chemotherapy after surgery

Exclusion Criteria:

* Have received anti-cancer therapy before surgery
* Have or had autoimmune disease in past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve (AUC) over the Dosing Interval at Cycle 1 | At the end of Cycle 1 (each cycle is 21 days)
  Defined as AUC calculated in Cycle 1 based on intensive PK assessment
Area Under the Concentration-time Curve (AUC) over the Dosing Interval at Cycle 6 | At the end of Cycle 6 (each cycle is 21 days)
  Defined as AUC calculated in Cycle 6 based on intensive PK assessment

SECONDARY OUTCOMES:
Disease-free Survival | From the date of randomization until the date of disease recurrence, occurrence of new primary NSCLC, or death of any cause, whichever occurs first, assessed up to Week 55
  Defined as the time from the date of randomization until the date of disease recurrence, occurrence of new primary NSCLC, or death of any cause, whichever occurs first.
Overall Survival | From the date of randomization until the date of death of any cause, assessed up to Week 55
  Defined as the time from the date of randomization until the date of death of any cause.

CONTACTS AND LOCATIONS:
Locations (24):
- Poland (2):
  - SB Investigative Site, Gdansk
  - SB Investigative Site, Otwock
- South Korea (14):
  - SB Investigative Site, Ansan
  - SB Investigative Site, Busan
  - SB Investigative Site, Daegu
  - SB Investigative Site, Hwasun
  - SB Investigative Site, Incheon
  - SB Investigative Site, Jinju
  - SB Investigative Site, Seongnam
  - SB Investigative Site 3, Seoul
  - SB Investigative Site 4, Seoul
  - SB Investigative Site 5, Seoul
  - SB Investigative Site 6, Seoul
  - SB Investigative Site 1, Suwon
  - SB Investigative Site 2, Suwon
  - SB Investigative Site, Ulsan
- Spain (3):
  - SB Investigative Site, A Coruña, Santiago de Compostela
  - SB Investigative Site, Jaén
  - SB Investigative Site, Málaga
- Turkey (Türkiye) (5):
  - SB Investigative Site, Adana
  - SB Investigative Site 1, Ankara
  - SB Investigative Site 2, Ankara
  - SB Investigative Site, Istanbul
  - SB Investigative Site, Izmir